CLINICAL TRIAL: NCT00057369
Title: Phase II, Randomized, Open-Label, Multi-Center Study to Evaluate the Safety and Efficacy of Dalbavancin Versus Vancomycin in the Treatment of Catheter-Related Bloodstream Infections With Suspected or Confirmed Gram-Positive Bacterial Pathogens
Brief Title: Safety and Efficacy of Dalbavancin Versus Vancomycin in the Treatment of Catheter-Related Bloodstream Infections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vicuron Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VER001-4
Record Dates: First submitted 2003-03-31; First posted 2003-04-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia | interventions — dalbavancin

INTERVENTIONS:
Drug: dalbavancin

SUMMARY:
This is a study to evaluate a new medication dosed once a week in the treatment of bacterial infections in the blood from intravenous catheters (CR-BSI). The primary objective is to evaluate the efficacy and safety of dalbavancin in the treatment of adults with CR-BSI relative to a standard of care treatment, vancomycin.

ELIGIBILITY:
* The patient or his/her legally authorized representative has given informed consent by means approved by the investigator's IRB/EC;
* > 18 years of age;
* Had one or more central venous catheters at the time initial signs of infection were evident;
* Creatinine clearance <50 mL/min;
* Bilirubin > 2x the upper limit of normal;
* Treatment with an antibiotic effective against Gram-positive bacterial infections for more than 24 hours within 48 hours of study medication initiation,
* Prolonged antibiotic therapy for CR-BSI anticipated (i.e., >2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88
Dates: Start 2001-02; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- Wellstar/Kennestone Hospital, Marietta, Georgia, United States

REFERENCES:
- [Derived] Gonzalez PL, Rappo U, Akinapelli K, McGregor JS, Puttagunta S, Dunne MW. Outcomes in Patients with Staphylococcus aureus Bacteremia Treated with Dalbavancin in Clinical Trials. Infect Dis Ther. 2022 Feb;11(1):423-434. doi: 10.1007/s40121-021-00568-7. Epub 2021 Dec 14. PMID 34905144